CLINICAL TRIAL: NCT04570800
Title: One Way to Diagnose Hepatic Insufficiency the First Postoperative Day After Resection: Prospective Cohort Study
Acronym: IGHI
Status: Completed | Type: Observational
Sponsor: Castilla-La Mancha Health Service (Other)
Responsible Party: Sponsor
Other Study IDs: VBG-IND-2014-01
Record Dates: First submitted 2020-09-25; First posted 2020-09-30 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Indocyanine Green; Postoperative Complications; Acute Liver Failure
Keywords: Indocyanine green; LIMON; Postoperative liver failure
MeSH Terms: conditions — Postoperative Complications; Liver Failure, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction: Hepatic insufficiency is a complication that puts the life of the patient undergoing resective surgery at risk. Thus, the diagnosis should be made early. The current gold standard allows its diagnosis on the fifth postoperative day.

Indocyanine green is a water soluble dye. When administered intravenously, it binds to plasma proteins and it is removed unchanged by bile, without experiencing enterohepatic recirculation, which allows estimating the function of hepatocytes and the function of hepato-splacnic flow. There is a measurement system named "Non-invasive liver function monitor" (LiMON®, PULSION Medical Systems, Munich, Germany), which allows the measurement of indocyanine green clearance at the patient's bedside.

Justification: The use of indocyanine green plasma disappearance during the perioperative period tries to know the exact value of the hepatic function in the most real conditions, when the excision has been performed, thus giving the investigators the actual value of the unresected liver. This allows te investigators to estimate the risk of hepatic insufficiency development that can lead to hepatic failure. Due to the characteristics of the test, it could get reliable results earlier than the current "gold standard " (50:50 Criteria on the 5th postoperative day).

Hypotheses and Objectives: The investigators hypothesized that the determination of the hepatic reserve by identifying the indocyanine plasma clearance in real time after hepatic parenchymal resection could lead to a more accurate and earlier statement of the hepatic reserve than current tests.

The aim of the study is to determine the usefulness of indocyanine green in the perioperative period to early diagnosis of hepatic failure.

Materials and Methods: A prospective observational post-authorization study (EPA-SP) is performed to study de usefulness of indocyanine green. The study was approved by the Ethics and Clinical Research Committee of the University General Hospital of Ciudad Real. Surgical patients scheduled for liver surgery, who agreed to be included in the study and signed an informed consent, were included in the study over a two-year period, after having understood the study objectives and its possible complications.

Measurements were performed with the LiMON® monitor prior to liver resection and on the first postoperative day to patients undergoing liver resection surgery and compared with gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Patients susceptible of receiving Surgical treatment
* Liver Disease with Surgical Indication
* Adulthood
* Accept Inclusion

Exclusion Criteria:

* History of Hypersensitivity to Indocyanine Green or Iodine
* Thyroid Pathology
* Underage Status
* Pregnant
* Irresectable Tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical patients scheduled for liver surgery, who agreed to be included in the study and signed the informed consent given to them following information given about the aims of the study and its possible complications, were included in the study consecutively for a period of two years
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Number of patients wich the plasma removal rate of Indocianin Green at 24h of surgery correlates with the existence of liver failure on the 5th postoperative day | 5 days
  Number of patients wich the plasma removal rate of Indocianin Green at 24h of surgery correlates with the existence of liver failure on the 5th postoperative day

SECONDARY OUTCOMES:
Number of patients wich the plasma removal rate of Indocianin Green at 24h of surgery correlates with the existence of liver failure on the 3th postoperative day | 3 days
  Number of patients the plasma removal rate of Indocianin Green at 24h of surgery correlates with the existence of liver failure on the 3th postoperative day